CLINICAL TRIAL: NCT02875171
Title: Assessment of Global Longitudinal Strain at Low Dose Anthracycline-based Chemotherapy for the Prediction of Subsequent Cardiotoxicity
Brief Title: Assessment of Global Longitudinal Strain for the Prediction of Anthracycline Induced Cardiotoxicity
Acronym: Anthracardio
Status: Completed | Type: Observational
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Clément Charbonnel, study principal investigator, Versailles Hospital
Other Study IDs: 11/17_Anthracardio
Record Dates: First submitted 2016-08-11; First posted 2016-08-23 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Cardiovascular Diseases
Keywords: Anthracyclines; Cardiotoxicity; 2-D Echocardiography
MeSH Terms: conditions — Cardiovascular Diseases; Cardiotoxicity | interventions — Anthracyclines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anthracycline therapy: Patients suffering from lymphoma or acute leukemia and requiring anthracycline administration were included
  Interventions: Drug: Anthracycline administration

INTERVENTIONS:
Drug: Anthracycline administration — Patients suffering from lymphoma or acute leukemia and requiring anthracycline administration were included
  Other Names: Anthracycline

SUMMARY:
Anthracycline therapy is well-known for its adverse cardiac effects. Anthracycline-induced cardiotoxicity (AIC) is associated with a poor prognosis; since classical heart failure treatment can potentially reverse cardiac dysfunction at the early stage of cardiac toxicity, early detection of AIC is crucial.

Transthoracic echocardiography is recommended for monitoring left ventricular function in patients receiving these molecules. In routine practice, left ventricular systolic function is mainly assessed by the left ventricular ejection fraction (LVEF), measured by two-dimensional echocardiography imaging. However, LVEF depends on the operator's experience and is not sensitive enough to detect subclinical myocardial dysfunction.

To overcome these limitations, two-dimensional speckle-tracking imaging has been proposed. This technique allows for a study of global and regional myocardial deformation, especially the longitudinal component, which appears to be the most sensitive one. Several studies have already emphasized the role of global longitudinal strain (GLS) to detect slight alterations in systolic function, especially in the setting of potentially cardiotoxic drugs and even after low to moderate doses of anthracyclines. A recent expert consensus paper strongly recommends GLS assessment for the detection of subclinical left ventricular dysfunction due to anthracycline therapy.

Although there is growing evidence that GLS can predict subsequent alterations in LVEF, few data exist on the optimal timing to perform echocardiography.

The investigators hypothesized that very early measurement of GLS in the time course of anthracycline therapy could predict subsequent left ventricular systolic dysfunction.

The aim of this study was, therefore, to determine whether assessment of GLS after 150 mg/m² of anthracyclines can predict AIC.

DETAILED DESCRIPTION:
Study population:

This is a single-centre, prospective cohort study. The patients are evaluated at four time points: visit 1 (V1), before the initiation of anthracycline therapy; visit 2 (V2), after reaching a cumulative dose of 150 mg/m²; visit 3 (V3), at the end of the treatment; and visit 4 (V4), 1 year after V1.

Clinical examination at each visit and standard echocardiography are performed. The study is approved by our ethics committee (EudraCT number 2011-002721- 22).

Two-dimensional echocardiography:

Echocardiography examinations are performed using a Vivid E9 imaging device (GE Medical systems, Horten, Norway). The left ventricular end-diastolic and endsystolic volumes are measured from the apical two- and four-chamber views; LVEF are calculated using Simpson's rule. GLS is computed from high frame rate (>50 frames per second) apical views (four-, two-, and three-chamber). By tracing the endocardial borders on an end-systolic frame, myocardial speckles are automatically tracked on the subsequent frames. Adequate tracking is verified, and manually corrected if necessary. GLS is obtained as the average of regional strains. Percentage change in GLS and absolute reduction in GLS are calculated between baseline and V2. Other classic diastolic and systolic parameters are recorded according to current guidelines. Digital loops are stored for off-line analysis. For LVEF and GLS, digital loops are done in triplicate to assess inter- and intraobserver variability. LVEF and GLS are analysed by two readers. The readers are blinded to each other's measurements and to the patient visit number.

Echocardiographic definition of AIC:

According to a recent consensus paper, anthracycline cardiotoxicity is defined as a decrease in the LVEF of >10 percentage points, to a value <53%, at V4. This decrease has to be confirmed by a repeat echocardiography performed a few weeks after V4.

ELIGIBILITY:
Inclusion Criteria:

1. patients suffering from lymphoma or leukemia and requiring anthracycline therapy;
2. over 18 years old;
3. baseline LVEF >50%.

Exclusion Criteria:

1. moderate to severe aortic or mitral valve disease;
2. pregnant or breastfeeding women;
3. atrial fibrillation;
4. very poor image quality defined by two or more myocardial segments inadequately visualized (17-segment model);
5. unstable cardiac condition such as pericardial effusion or acute coronary syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from lymphoma or acute leukemia and requiring anthracycline administration were included
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2011-10; Primary Completion 2015-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Dynamic changes in Global Longitudinal Strain (GLS) throughout the visits | 1 year
  Determine whether assessment of GLS after 150 mg/m² of anthracyclines can predict AIC.

CONTACTS AND LOCATIONS:
Overall Officials: Charbonnel Clément, MD, Principal Investigator — CH Versailles
Locations (1):
- CH Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No